CLINICAL TRIAL: NCT01017939
Title: An Abiraterone Acetate Plus Prednisone Drug-Drug Interaction Study With Dextromethorphan and Theophylline in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Drug-Drug Interaction Study of Abiraterone Acetate Plus Prednisone With Dextromethorphan and Theophylline in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017128; COU-AA-015 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Metastatic castration resistant prostate cancer; Metastatic castration refractory prostate cancer; Prostate cancer; Abiraterone acetate; CB7630
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Dextromethorphan; Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: abiraterone + prednisone + dextromethorphan (Experimental): Group A will assess the effect of multiple doses of abiraterone acetate plus prednisone on CYP2D6 using 2 single doses of dextromethorphan hydrobromide as a probe drug.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: Dextromethorphan hydrobromide
- Group B: abiraterone + prednisone + theophylline (Experimental): Group B will assess the effect of multiple doses of abiraterone acetate plus prednisone on CYP1A2 using 2 single doses of theophylline as a probe drug.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: Theophylline

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate 1000 mg tablets administered orally once daily beginning on Cycle 1 Day 1 up to the time of disease progression
Drug: Prednisone — Prednisone 5mg tablets administered orally twice daily beginning on Cycle 1 Day 1 up to the time of disease progression
Drug: Dextromethorphan hydrobromide — Dextromethorphan hydrobromide 30 mg capsules administered orally on Cycle 1 Day -8 and Cycle 1 Day 8 under fasting conditions
  Arms: Group A: abiraterone + prednisone + dextromethorphan
Drug: Theophylline — Theophylline 100 mg tablets administered orally on Cycle 1 Day -8 and Cycle 1 Day 8 under fasting conditions
  Arms: Group B: abiraterone + prednisone + theophylline

SUMMARY:
The purpose of this study is to evaluate the effects of multiple doses of abiraterone acetate plus prednisone on the pharmacokinetics (study of what the body does to a drug) of single doses of dextromethorphan hydrobromide and theophylline in patients with castration resistant prostate cancer.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study of abiraterone acetate plus prednisone in male patients with metastatic castration-resistant prostate cancer. This study will consist of screening, treatment, and follow-up periods, and will have 2 study groups. Patients in Group A and B will receive daily abiraterone acetate (1000 mg) plus prednisone (5 mg) twice daily beginning on Cycle 1 Day 1 until disease progression. Patients in Group A will take dextromethorphan hydrobromide 30 mg administered orally once daily on Day -8 and Day 8 of Cycle 1. Patients in Group B will take theophylline 100 mg administered orally once daily on Day -8 and Day 8 of Cycle 1. Serial pharmacokinetic samples will be collected and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Documented metastatic disease
* Documented prostate specific antigen (PSA) progression according to Prostate Cancer Working Group 2 criteria, with PSA value >=2 ng/mL despite medical or surgical castration, or prostate cancer progression documented by radiographic progression according to Response Evaluation Criteria In Solid Tumors criteria
* Surgically or medically castrated with testosterone levels of <50 ng/dL
* Eastern Cooperative Oncology Group (ECOG) Performance Status of <=2
* Group A only: genomic testing at screening indicating CYP2D6 extensive metabolizer status
* Protocol-defined laboratory values

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Group A only: genomic testing at screening indicating CYP2D6 non-extensive metabolizer status, or prior treatment with dextromethorphan-containing medication or any medication that is a strong inhibitor or inducer of CYP2D6 within 5 half-lives of that drug or 7 days, whichever is longer, prior to Cycle 1 Day -8
* Group B only: prior treatment with theophylline or any medication that is a strong inhibitor or inducer of CYP1A2 within 5 half-lives of that drug or 7 days, whichever is longer, prior to Cycle 1 Day -8
* Abnormal liver function
* Uncontrolled hypertension (repeated systolic blood pressure >=160 mmHg, or diastolic blood pressure >=95 mmHg)
* Active or symptomatic viral hepatitis or chronic liver disease
* Known brain metastasis
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association Class III or IV heart disease or cardiac ejection fraction measurement of <50% at baseline
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
* Surgery or local prostatic intervention within 28 days of the first dose, and any clinically relevant sequelae from the surgery must have resolved prior to Cycle 1 Day 1
* Radiotherapy or immunotherapy within 28 days, or single fraction of palliative radiotherapy within 14 days of administration of Cycle 1 Day 1
* Any acute toxicities due to prior therapy that have not resolved
* Current enrollment in an investigational drug or device study or participation in such a study within 28 days of Cycle 1 Day 1
* Previous abiraterone acetate or other investigational CYP17 inhibitor (eg, TAK-700)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ratio of the mean area under the concentration curve (AUC) of dextromethorphan, dextrorphan, and parent/metabolite, with and without co-administration of abiraterone acetate and prednisone | Cycle 1 Day -8 and Day 8
Ratio of the mean maximum plasma concentration (Cmax) of dextromethorphan, dextrorphan, and parent/metabolite, with and without co-administration of abiraterone acetate and prednisone | Cycle 1 Day -8 and Day 8
Ratio of the mean area under the concentration curve (AUC) of theophylline with and without co-administration of abiraterone acetate and prednisone | Cycle 1 Day -8 and Day 8
Ratio of the mean maximum plasma concentration (Cmax) of theophylline with and without co-administration of abiraterone acetate and prednisone | Cycle 1 Day -8 and Day 8

SECONDARY OUTCOMES:
Number of participants reporting adverse events | Up to 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- United States (4):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Beverly Hills, California
  - START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - San Antonio, Texas
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Vancouver, British Columbia

REFERENCES:
- See also: An Abiraterone Acetate Plus Prednisone Drug-Drug Interaction Study with Dextromethorphan and Theophylline in Patients with Metastatic Castration-Resistant Prostate Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2416&filename=CR017128_CSR.pdf